CLINICAL TRIAL: NCT01656382
Title: Safety, Efficacy, and Pharmacokinetics of Amphotericin B Lipid Complex at 10 mg/kg/d for 7 Days or 5.0 mg/kg/d for 14 Days as Induction Therapy for Disseminated Cryptococcosis in Patients With HIV
Brief Title: Safety, Efficacy, and Pharmacokinetics of Amphotericin B Lipid Complex
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-273
Record Dates: First submitted 2007-04-24; First posted 2012-08-03 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Invasive Cryptococcosis
Keywords: ABLC; cryptococcosis
MeSH Terms: conditions — Cryptococcosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 mg/kg/d ABLC x 14 days (Active Comparator): 5 mg/kg/d of Amphotericin B Lipid Complex for 14 days
  Interventions: Drug: ABLC
- 10/kg/kg/d x 7 days (Experimental): 10 mg/kg/d of Amphotericin B Lipid Complex for 7 days
  Interventions: Drug: ABLC

INTERVENTIONS:
Drug: ABLC

SUMMARY:
The purpose of this study is to determine if initial therapy with ABLC at 10/mg/kg/d for 7 days are at least effective as ABLC at 5.0 mg/kg/d X 14 days as induction treatment of patients with disseminated cryptococcosis and HIV.

DETAILED DESCRIPTION:
This is a randomized, open label, prospective study of ABLC at 5.0 and 10.0 mg/kg/d for treatment of patients with cryptococcal meningitis. Patients will be randomly assigned in a 1:1 ratio to receive 5.0 or 10.0 mg/kg/d of ABLC as induction therapy for cryptococcal meningitis. Patients receiving 10 mg/kg/d doses will be treated with ABLC for 7 days whereas patients receiving ABLC at 5.0 mg/kg/d will receive 14 days of ABLC therapy. After completion of induction therapy subjects will receive long-term fluconazole maintenance therapy at the discretion of the treating physician. The study will be conducted at the Washington Hospital Center

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cryptococcal meningitis based on any of the following:

   * Cerebrospinal fluid positive for C. neoformans
   * Cerebrospinal fluid positive for cryptococcal antigen
2. Male or female 18 years of age or older.
3. All female patients must be non-lactating and have a negative serum pregnancy test at time of screening. Females of childbearing potential must be using a medically acceptable method of contraception and agree to continue its use during the study period, or must be one year postmenopausal, or have been surgically sterilized.
4. Willing and able to give a signed informed consent, or have a legally authorized representative who is willing or able to give consent

Exclusion Criteria:

1. A history or evidence of hypersensitivity to AmB or any of its metabolites.
2. A history or evidence of any psychiatric, neurological metabolic, or other chronic condition, which in the investigator's opinion, would make the patient unsuitable for the study or interfere with the evaluation of ABLC.
3. Inability to comply with the procedures of the study.
4. Patients who have received greater than 72 hours of therapy with another systemic antifungal agent within 2 weeks prior to enrollment
5. Patients with any of the following abnormal laboratory values

   * Baseline creatinine clearance of less than 50.
   * Bilirubin of greater than 5 times the upper limit of normal
   * AST or ALT of greater than 10 times the upper limit of normal
6. Life expectancy of less than 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Survival
Time to Sterilization of CSF

SECONDARY OUTCOMES:
Infusion related and renal toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Shoham, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States